CLINICAL TRIAL: NCT06071468
Title: Registry of the Patient Experience for Carpal Tunnel Release (MISSION)
Brief Title: Registry of the Patient Experience for Carpal Tunnel Release
Acronym: MISSION
Status: Active, not recruiting | Type: Observational
Sponsor: Sonex Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 90154-TP
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Carpal Tunnel Syndrome; CTS
Keywords: Ultrasound Guided Carpal Tunnel Release; CTR-US; ECTR; OCTR
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Ultrasound Guided Carpal Tunnel Release (CTR-US): Carpal Tunnel Release using CTR-US technique
  Interventions: Device: UltraGuideCTR (Device) with Ultrasound Guided Carpal Tunnel Release (CTR-US)
- Open Carpal Tunnel Release (OCTR): Carpal Tunnel Release Using Open Carpal Tunnel Release (OCTR)
  Interventions: Procedure: Open CTR
- Endoscopic Carpal Tunnel Release (ECTR): Carpal Tunnel Release Using Endoscopic Carpal Tunnel Release (ECTR)
  Interventions: Procedure: Endocscopic CTR

INTERVENTIONS:
Device: UltraGuideCTR (Device) with Ultrasound Guided Carpal Tunnel Release (CTR-US) — The UltraGuideCTR is a commercially available medical device specifically developed to facilitate CTR-US. The device is a single-use, hand-held device that is inserted into the carpal tunnel through a small (typically < 5 mm) wrist incision using continuous US guidance. The working tip of the UltraGuideCTR consists of two inflatable balloons that border a centrally located, retractable retrograde cutting knife. When inflated with sterile saline, the balloons increase the diameter of the tip from 4 mm to 8 mm. After the tip is positioned within the transverse safe zone of the carpal tunnel, the balloons are inflated to create space in the carpal tunnel, the blade is activated, and the TCL is transected in a retrograde manner. Following TCL transection, the blade is recessed, the balloons deflated, and the device is removed. The TCL is probed to ensure a complete release. The entire procedure is performed using US guidance.
  Groups: Ultrasound Guided Carpal Tunnel Release (CTR-US)
Procedure: Endocscopic CTR — Endoscopic CTR makes one or two short incisions to introduce instruments for visualizing. The key procedural steps involved in Endoscopic CTR are listed below.
  1. Following the delivery of anesthesia, the surgeon makes a small wrist incision (usually less than 1.5 cm), with or without a small palmar incision (usually less than 1.5 cm, depending on whether they are using a single portal or double portal technique, respectively.
  2. A series of dilators and raspers are used to create space in the carpal tunnel and clear synovial tissue from the undersurface fo the TCL.
  3. A camera attached to a narrow tube (endoscope) is inserted into the carpal tunnel.
  4. The transverse carpal ligament (which forms the roof of the carpal tunnel) is identified.
  5. Using specialized cutting instruments and endoscopic guidance, the surgeon transects the TCL.
  6. Endoscopic visualization and/or probing are used to confirm a complete release.
  7. The wound(s) is/are typically closed with sutures.
  Other Names: ECTR
  Groups: Endoscopic Carpal Tunnel Release (ECTR)
Procedure: Open CTR — OCTR is the most commonly used CTR technique in the United States.The key procedural steps involved in OCTR are listed below.
  1. Following the delivery of anesthesia, an incision is made in the palm directly over the carpal tunnel.
  2. The surgeon cuts through the palmar fascia to identify the TCL.
  3. The surgeon transects the TCL with a scalpel and/or similar cutting instruments.
  4. The surgeon inspects the carpal tunnel to ensure proper decompression.
  5. The wound is closed with sutures.
  Other Names: OCTR
  Groups: Open Carpal Tunnel Release (OCTR)

SUMMARY:
Multi-center study to collect large scale, multidimensional real-world data on patients undergoing carpal tunnel release (CTR).

DETAILED DESCRIPTION:
Multicenter prospective Registry of patients with symptomatic carpal tunnel syndrome (CTS) treated (unilateral or simultaneous bilateral) by Ultrasound guided CTR (CTR-US), Endoscopic CTR (ECTR), or Open CTR (OCTR).

ELIGIBILITY:
Inclusion Criteria 1. ≥18 years of age 2. Clinical diagnosis of unilateral or bilateral CTS 3. A clinical decision has been made to perform CTR on one or both hands 4. CTS-6 score ≥12 in the target hand(s)* 5. Confirmatory diagnostic testing in the target hand(s)*:

1. CTR-US: Confirmatory diagnostic testing with ultrasound (median nerve cross-sectional area ≥10 mm2 in the proximal carpal tunnel region)
2. ECTR or OCTR: Confirmatory electrodiagnostic testing 6. Prior failure of one or more nonsurgical treatment options (e.g., physical activity modification, bracing, splinting, corticosteroid injection) in the target hand(s) 7. Patient agrees to complete follow-up questionnaires over a 24-month period 8. Patient has a valid smart phone number and/or email address to receive and answer follow-up questionnaires

Note: An asterisk (*) denotes that this criterion must be applied to the target hand for unilateral CTR procedures, or to both hands for simultaneous bilateral CTR procedures.

Exclusion Criteria:

1. Patient meets any of the contraindications per Instruction For Use (IFU)
2. Patient has other medical, social, or psychological conditions that, in the opinion of the investigator, preclude them from completing all registry requirements.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Carpal Tunnel Syndrome meeting study eligibility criteria. Patients are invited to volunteer to participate at selected study sites.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire - Symptom Severity Scale (BCTQ-SSS) | 24 Months
  Scoring for the BCTQ- SSS ranges from 1 to 5, with higher scores indicating more severe symptoms, and is calculated as the mean of each response. The change in BCTQ-SSS score at the 24-month follow-up relative to baseline.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire - Functional Status Scale (BCTQ-FSS) | 24 Months
  Scoring for the BCTQ-FSS ranges from 1 to 5, with higher scores indicating more functional limitation, and is calculated as the mean of each response. The change in BCTQ-FSS score at the 24-month follow-up relative to baseline.
Numeric Pain Scale | 24 Months
  Subjects will be asked to rate their wrist pain severity on a scale of 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain". The change in Numeric Pain Scale score at the 24-month follow-up relative to baseline.
EuroQoL 5-Dimension 5-Level (EQ-5D-5L) | 24 Months
  The EQ-5D-5L measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking consisting of: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The change in EQ-5D-5L score at the 24-month follow-up relative to baseline.
Device and/or Procedure Related Adverse Events | 24 Months
  Incidence of device- or procedure-related AEs within 24 months of treatment.
Global Satisfaction with Carpal Tunnel Release Procedure | 24 Months
  Subjects will be asked to rate their satisfaction with the carpal tunnel release procedure and how likely they are to recommend their carpal tunnel release procedure to a friend or colleague on a scale from 0-10 with 0 being not at all likely and 10 being extremely likely. Satisfaction will be reported with the following options: Very Satisfied, Satisfied, Neither Satisfied or dissatisfied, Dissatisfied or Very dissatisfied.

OTHER OUTCOMES:
Pain medication use through 24 months | 24 Months
  Post-index procedure use of pain medication by type (prescription [Tramadol (Ultram) or tapentadol (Nucynta) vs other prescribed opioids / narcotics], non-prescription)
Additional surgical interventions through 24 months | 24 Months
  * Post-index CTR revision surgery by type (e.g., CTR-US, ECTR, OCTR, other) and reason (e.g., persistent symptoms, recurrent symptoms)
  * Other post-index CTR surgery by side and surgery type (e.g., CTR, trigger finger release, trigger thumb release, release for De Quervain's syndrome, cubital tunnel

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Marwin, MD, MBA, Principal Investigator — Bluegrass Orthopaedics
Locations (33):
- United States (33):
  - The Orthopaedic Group P.C. (CTR-US), Foley, Alabama
  - Phoenix Hand (CTR-US), Scottsdale, Arizona
  - Orthopaedics Associates of Hartford (OCTR), Glastonbury, Connecticut
  - Aventura Hand Center (CTR-US), Aventura, Florida
  - Orthopaedic Associates (CTR-US), Fort Walton Beach, Florida
  - Central Florida Orthopaedic Surgery Associates, P.L (CTR-US), Lakeland, Florida
  - Melbourne Hand Center (OCTR), Melbourne, Florida
  - Miami Hand Center (NHVP), Miami, Florida
  - The Orthopaedic Hand and Arm Center (CTR-US), Miami Lakes, Florida
  - Tri-State Orthopaedics (CTR-US), Evansville, Indiana
  - Bluegrass Orthopaedics (CTR-US), Lexington, Kentucky
  - Cape Cod Orthopaedics (CTR-US), Hyannis, Massachusetts
  - Excel Orthopaedic Specialists (CTR-US), Woburn, Massachusetts
  - Mendelson Orthopedic PC (CTR-US), Troy, Michigan
  - Twin Cities Orthopedics (OCTR), Edina, Minnesota
  - Mississippi Sports Medicine& Orthopedic Center (ECTR), Jackson, Mississippi
  - Orthopedic Asociates (CTR-US), St Louis, Missouri
  - Hand Center of Nevada (CTR-US), Las Vegas, Nevada
  - Dartmouth Hitchcock Clinic (ECTR), Lebanon, New Hampshire
  - Mobility Bone and Joint Institute (CTR-US), Salem, New Hampshire
  - New Mexico Orthopedics (CTR-US), Albuquerque, New Mexico
  - Buffalo Surgery Center (CTR-US), Amherst, New York
  - The Bone&Joint Surgery Clinic (CTR-US), Raleigh, North Carolina
  - The Center (ECTR), Bend, Oregon
  - Slocum Research & Education Foundation (ECTR), Eugene, Oregon
  - Meadville Medical Center (ECTR), Meadville, Pennsylvania
  - University Orthopedics Center (OCTR), State College, Pennsylvania
  - University Orthopedics, Inc.(OCTR), East Providence, Rhode Island
  - Ortho SC (CTR-US), Conway, South Carolina
  - Prisma Health (ECTR), Greenville, South Carolina
  - Sports Orthopedics & Spine (CTR-US), Jackson, Tennessee
  - North Texas Hand Center (CTR-US), Denton, Texas
  - North Texas Orthopedics and Spine Center (CTR-US), Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
This study is privately funded and IPD will not be available for use beyond the study Sponsor or the participating Investigational Sites.